CLINICAL TRIAL: NCT05601869
Title: Impact of Improving Footwear Options for Women Veterans With Amputations
Brief Title: Impact of Improving Footwear Options
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: D4256-R
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Amputation
Keywords: Artificial Limbs; Amputation; Leg Prosthesis; Body Image; Community Participation; Social Participation

STUDY DESIGN:
Intervention Model Description: Pretest-Posttest Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Participants in this arm receive a new prosthesis system designed to improve footwear options.
  Interventions: Device: RECOVER Prosthetic Ankle-Feet System

INTERVENTIONS:
Device: RECOVER Prosthetic Ankle-Feet System — The RECOVER prosthetic ankle-feet system includes a single prosthetic ankle joint that can be easily attached to 3D printed feet. The feet are designed to fit specifically within different footwear.
  Other Names: RECOVER AFS

SUMMARY:
Veterans with leg amputations have limited footwear options because their artificial feet do not change shapes for different shoes. Studies have shown that women with amputations receive more frequent prosthetics care than men, but are less satisfied with the fit, comfort, and appearance of their prostheses. The investigators' previous research indicates that women Veterans would like to be able to wear a broader variety of footwear, and those who perceive more footwear limitations tend to have poorer body image and community participation. A new prosthesis designed by the investigators' group allows Veterans with amputations to use their footwear of choice using 3D-printed artificial feet with a single ankle. The novel prosthesis will be tested in this project with women Veterans with amputations to determine the impact of improving footwear options on body image and community participation.

DETAILED DESCRIPTION:
Background - Veterans with leg amputations have limited footwear options because their artificial feet do not change shapes for different shoes. Studies have shown that women with amputations receive more frequent prosthetics care than men, but are less satisfied with the fit, comfort, and appearance of their prostheses. The investigators' previous research indicates that women Veterans would like to be able to wear a broader variety of footwear, and those who perceive more footwear limitations tend to have poorer body image and community participation. A new prosthesis designed by the investigators' group allows Veterans with amputations to use their footwear of choice using 3D-printed artificial feet with a single ankle. The investigators seek to understand the impact of improving footwear options for women Veterans with amputations on body image and community participation following a 6-month take-home trial.

Research Questions (Objectives) - The purpose of this project is to evaluate the effect of a new prosthetic ankle-feet system on body image and participation among women Veterans with lower limb amputations.

Relevance to VA - Women Veterans with amputations is a small but growing demographic of US military Veterans. Women with amputations receive more frequent prosthetics care, but are less satisfied with the fit, comfort, and appearance of their prostheses than men. These findings are not surprising as most prosthesis components are not gender-specific and seem to have been designed for men. The investigators' group has developed a 3D-printed ankle feet system customized to fit a wide range of footwear, including shoes of different heel heights and widths. This new prosthesis system dramatically improves footwear options for persons using leg prostheses, enabling potential to increase body image and community participation for women Veterans with leg amputations. This study is an important next step in the investigators' line of research and is needed to determine the impact of improving footwear options for this important and growing subpopulation of Veterans.

Number of Research Participants (Sample Size) - We will recruit up to 18 women Veterans with transtibial amputations to participate and anticipate that at least 12 participants will complete the entire study. The investigators plan to screen women Veterans from a national sample to accomplish the recruitment and completion goals.

Participating Sites - Minneapolis VA Health Care System

Duration of Participant Intake (Study Duration) - This project is projected to occur over three years. The project will begin with a 6-month start-up period and recruitment will continue for two years following start-up. Recruitment will conclude with 6-months remaining in the study timeline, which will be used for dissemination of results and closure of the project.

Treatment (follow-up) - The intervention being tested is a new prosthetic ankle-feet prosthesis that women Veterans will wear for 6-months in their home and community environments. The investigators will follow-up with participants after 1-month and after 6-months of home and community use.

Endpoints - The primary outcomes for this study are body image (Amputee-specific Body Image Scale - Revised) and ability to participate in social roles and activities (PROMIS - Ability to Participate in Social Roles and Activities).

Qualitative Data - In addition to measuring body image and participation, the investigators will conduct semi-structured interviews will participants to develop further understanding of the benefits and drawbacks of using the new prosthetic ankle-feet system. Participants will also complete a photovoice task in which they will be asked to take photos regarding their experience using the new prosthetic ankle-feet system. These photos will then be used as talking points during the semi-structured interview to improve the understanding of the user experience with the system.

ELIGIBILITY:
Inclusion Criteria:

* US military Veterans that identify as women
* Transtibial (below-knee) amputation
* Using a definitive prosthesis for at least 6 months (limb has accommodated to prosthesis use post-amputation)
* Well fitting and well aligned prosthesis
* Blessed Orientation-Memory-Concentration (Short Blessed) score between 0-6
* Access to computer, tablet, or smart phone and internet for video conferencing and RedCap data collection

Exclusion Criteria:

* Residual limb skin problems
* Residual limb too long to accommodate the RECOVER prosthetic ankle-feet system
* Unable or unwilling to travel to Minneapolis
* Not a regular prosthesis user
* Mass over 125 kg
* Documented neurocognitive disorder (e.g., dementia) with evidence of impact on activities of daily living and/or instrumental activities of daily living
* Baseline ABIS-R or PROMIS-APSRA scores at the maximum levels (no room for improvement on primary outcomes)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This project focuses on Veterans identifying as women.
Enrollment: 18 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Amputation-Specific Body Image Scale-Revised (ABIS-R) Change | Baseline, 1-month, 6-months
  The ABIS-R is a 14-item scale that assesses body image disturbance among individuals with amputations. Responses are reported on a 1 to 3 scale, with higher values representing greater body image disturbance.
PROMIS Ability to Participate in Social Roles and Activities (PROMIS APSRA) Change | Baseline, 1-month, 6-months
  The PROMIS Ability to Participate in Social Roles and Activities (PROMIS-APSRA) specifically measures one's ability to participate in social roles and activities, including one's ability to do leisure activities and activities with friends and family. The PROMISAPSRA is an 8-item form that uses a 5-point scale, where higher values indicate a higher degree of ability to participate.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H Hansen, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No